CLINICAL TRIAL: NCT06858709
Title: Effect of Adding Electroacupuncture Combined With Standard Anti Chemotherapy-induced Peripheral Neuropathy Drugs to Anti-cancer Therapy-induced Peripheral Neuropathy: a Randomized Multicentered Clinical Trial.
Brief Title: Effect of Adding Electroacupuncture to Anti-cancer Therapy-induced Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZNYYKL2025013
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN); Cancer
Keywords: Chemotherapy-induced peripheral neuropathy (CIPN); electroacupuncture treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- True acupuncture + standard anti chemotherapy-induced peripheral neuropathy treatment (Experimental)
  Interventions: Procedure: True acupuncture + standard anti chemotherapy-induced peripheral neuropathy treatment
- Sham acupuncture +standard anti chemotherapy-induced peripheral neuropathy treatment (Placebo Comparator)
  Interventions: Procedure: Sham acupuncture +standard anti chemotherapy-induced peripheral neuropathy treatment

INTERVENTIONS:
Procedure: True acupuncture + standard anti chemotherapy-induced peripheral neuropathy treatment — Participants will receive a total of 8 treatments over 6 weeks, with twice a week treatments for the first and the forth weeks and weekly treatment for the remaining weeks.The acupuncturists will insert needles into the acupoints and manipulate the needles until"de qi"sensation is achieved and reported by the participants. In the meantime, participants will receive the same standard anti-CIPN treatments.
  Arms: True acupuncture + standard anti chemotherapy-induced peripheral neuropathy treatment
Procedure: Sham acupuncture +standard anti chemotherapy-induced peripheral neuropathy treatment — The sham acupuncture comprised a core standardized prescription of minimally invasive, shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive minimal acupuncture treatment without electrical stimulation at the same time as the intervention group. Care was taken to avoid "de qi" sensation. In the meantime, participants will receive the same standard anti-CIPN treatments.
  Arms: Sham acupuncture +standard anti chemotherapy-induced peripheral neuropathy treatment

SUMMARY:
This study is being done to evaluate the potential benefits of using electroacupuncture to reduce the severity of chemotherapy-induced peripheral neuropathy for patients with peripheral neuropathy after chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) refers to symptoms caused by chemotherapy drugs, such as numbness, tingling sensation, decreased sensation, hypersensitivity, or even limb dysfunction and muscle atrophy, which can be divided into five grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). The higher the grade, the more severe the symptoms. The incidence of chemotherapy-induced peripheral neuropathy (CIPN) reached 68.1% within the first month after treatment. About one-third of patients may develop chronic CIPN six months or more after chemotherapy, which significantly impairs the patients' quality of life. Electroacupuncture, as a nonpharmacologic therapy, is minimally invasive, with few side effects, and has demonstrated efficacy in various conditions including chemotherapy-induced nausea and vomiting. However, studies on its effectiveness against CIPN still yields inconsistent results.

This is a parallel-group, double-blinded (participants and statisticians), randomized controlled study that investigates the role of electroacupuncture compared with sham acupuncture for patients receiving chemotherapy. Both groups will receive the standard therapy for CIPN. On this basis, electroacupuncture or sham acupuncture will be randomly administered to the two groups. The investigators will explore the efficiency of electroacupuncture in reducing the severity of CIPN. Primary and secondary outcomes and adverse events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, of any nationality.
* Patients diagnosed with malignant tumor.
* Eligible patients will report altered sensations and/or pain and/or other neurological symptoms, with a grade between 2-3 for chemotherapy-induced peripheral neuropathy on the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events-version 5.0 (NCI-CTCAE.v-5.0).
* Predicted life expectancy of ≥3 months.
* Intact skin without any breaches or purulent discharge.
* Written informed consent by the patient before enrolment Patients must be able to comply with the study protocol, which includes attending the treatment sessions on time and completing the study questionnaires in accordance with the study protocol.

Exclusion Criteria:

* History of pre-existing peripheral neuropathy before chemotherapy, including alcoholism, vitamin B deficiency, diabetes, HIV, congenital neuropathy, and toxic neuropathy.
* Patients with skin damage, pus or scar at the acupuncture stimulation area.
* Patients who are pregnant or breastfeeding.
* Significant mental conditions.
* Patients not fulfilling the inclusion criteria.
* Patients receiving other acupuncture treatments during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference of the CIPN grade from baseline to week 6 after baseline | From enrollment to week 6
  The primary outcome will be the proportion of patients whose CIPN grade improved after the completion of 8 acupuncture treatments sessions.

SECONDARY OUTCOMES:
Changes in FACT/NTX subscale baseline to 6 weeks | baseline,week 3, week6
  Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) is a 38-item self-reported questionnaire: the 27-item general assessment of Quality of Life scale (FACT-G),alongside its 11-item neurotoxicity-specific module. Considering the patient's compliance, the investigators only require the patient to complete the 11-item neurotoxicity-specific module.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No